CLINICAL TRIAL: NCT06930937
Title: An Open Label, Randomized, Four-period, Twotreatment, Two-sequence, Fully Replicate, Crossover, Balanced, Single Dose Oral Bioequivalence Study
Brief Title: To Compare and Evaluate the Oral Bioavailability of Edoxaban 60 mg Film Coated Tablet With That of Lixiana® 60 mg Filmtabletten (Film Coated Tablet) (Edoxaban) in Healthy, Adult, Human Subjects Under Fasting Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Humanis Saglık Anonim Sirketi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: Protocol No.: C1B03118
Record Dates: First submitted 2025-04-09; First posted 2025-04-16 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2024-11

CONDITIONS: Prevention of Stroke or Systemic Embolism; Deep Vein Thrombosis (DVT); Pulmonary Embolism (PE)
MeSH Terms: conditions — Venous Thrombosis; Pulmonary Embolism | interventions — edoxaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Edoxaban Film Coated Tablet (Experimental): Edoxaban Film Coated Tablet (60 mg)
  Interventions: Other: Lixiana® Film Coated Tablet; Other: Edoxaban Film Coated Tablet
- Lixiana® filmtabletten (Film Coated Tablet) (Edoxaban) (Active Comparator)
  Interventions: Other: Lixiana® Film Coated Tablet; Other: Edoxaban Film Coated Tablet

INTERVENTIONS:
Other: Lixiana® Film Coated Tablet — Lixiana® 60 mg filmtabletten (Film Coated Tablet) (Edoxaban)
Other: Edoxaban Film Coated Tablet — Edoxaban 60 mg Film Coated Tablet

SUMMARY:
* To compare and evaluate the oral bioavailability of Edoxaban 60 mg Film Coated Tablet with that of Lixiana® 60 mg filmtabletten (Film Coated Tablet (Edoxaban) in healthy, adult, human subjects under fasting conditions.
* To monitor the safety and tolerability of the subjects.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 55 years old, both inclusive.
* Gender: Male and/or non-pregnant, non-lactating female.

A. Female of child-bearing potential had a negative serum beta human chorionic gonadotropin (β HCG) pregnancy test performed within 28 days prior to first dosing day. They used an acceptable form of contraception. For female of child-bearing potential, acceptable forms of contraception included the following:

i. Non hormonal intrauterine device in place for at least 3 months prior to the start of the study and remaining in place during the study period, or ii. Barrier methods containing or used in conjunction with a spermicidal agent, or iii. Surgical sterilization or iv. Practicing sexual abstinence throughout the course of the study.

B. Female was not considered of child-bearing potential if one of the following was reported and documented on the medical history:

i. Postmenopausal with spontaneous amenorrhea for at least one year, or ii. Spontaneous amenorrhea for more than 6 months and less than one year with Serum Follicular Stimulating Hormone (FSH) level > 40 mIU/mL, or iii. Bilateral oophorectomy with or without a hysterectomy and an absence of bleeding for at least 6 months, or iv. Total hysterectomy and an absence of bleeding for at least 3 months.

* BMI: 18.5 to 30.0 kg/m2, both inclusive; BMI value was rounded off to one significant digit after decimal point (e.g. 30.04 rounds down to 30.0, while 18.45 rounds up to 18.5).
* Volunteers had a body weight of more than 60 kg
* Non-smokers and non-tobacco users (i.e. had no past history of smoking and tobacco consuming for at least one year prior to study).
* Able to communicate effectively with study personnel.
* Willing to provide written informed consent to participate in the study.
* All volunteers were judged by the principal or sub-investigator or physician as normal and healthy during a pre-study safety assessment performed within 28 days of the first dose of study medication which will include:

  1. A physical examination (clinical examination) with no clinically significant finding.

Exclusion Criteria

* History of allergic responses to Edoxaban or other related drugs, or any of its formulation ingredients.
* Had significant diseases or clinically significant abnormal findings during screening [medical history, physical examination (clinical examination), laboratory evaluations, ECG recording, gynecological history and examination (including pelvic examination and routine breast examination) (for female volunteers)].
* Any disease or condition like diabetes, psychosis or others, which might compromise the haemopoietic, gastrointestinal, renal, hepatic, cardiovascular, respiratory, central nervous system or any other body system.
* History or presence of bronchial asthma.
* Used any hormone replacement therapy within 3 months prior to the first dose of study medication.
* Used any depot injection or implant of any drug within 3 months prior to the first dose of study medication.
* Used CYP enzyme inhibitors or inducers within 30 days prior to the first dose of study medication (see https://drug-interactions.medicine.iu.edu/MainTable.aspx).
* History or evidence of drug dependence or of alcoholism or of moderate alcohol use.
* History of difficulty with donating blood or difficulty in accessibility of veins.
* A positive hepatitis screen (includes subtypes B & C).
* A positive test result for HIV antibody.
* Volunteers who had received a known investigational drug within seven elimination half-life of the administered drug prior to the first dose of study medication.
* Volunteers who had donated blood or loss of blood 50 ml to 100 ml within 30 days or 101 ml to 200 ml within 60 days or >200 ml within 90 days (excluding volume drawn at screening for this study) prior to first dose of study medication, whichever was greater.
* History of difficulty in swallowing or of any gastrointestinal disease, which could affect drug absorption.
* Intolerance to venipuncture
* Any food allergy, intolerance, restriction or special diet that, in the opinion of the principal investigator or sub-investigator, could contraindicate the volunteer's participation in this study.
* Institutionalized volunteers.
* Used any prescribed medications [including aspirin and other antiplatelet agents, antithrombotic agents, fibrinolytic therapy, nonsteroidal anti-inflammatory drugs (NSAIDs), selective serotonin reuptake inhibitors and serotonin-norepinephrine reuptake inhibitors] within 14 days prior to the first dose of study medication.
* Used any OTC products, vitamin and herbal products, etc., within 7 days prior to the first dose of study medication.
* Used grapefruit and grapefruit containing products within 7 days prior to the first dose of study medication.
* Ingestion of any caffeine or xanthine products (i.e. coffee, tea, chocolate, and caffeine-containing sodas, colas, etc.), recreational drugs, alcohol or other alcohol containing products within 48 hours prior to the first dose of study medication.
* Ingestion of any unusual diet, for whatever reason (e.g.: low sodium) for three weeks prior to the first dose of study medication.
* Volunteer had a platelet count below the lower limit of the normal range during screening.
* Volunteer had an INR and Prothrombin Time and/or Activated Partial Thromboplastin Time value higher than 1.1 times of the upper limit of normal ranges during screening.
* Volunteers had SGPT, SGOT and alkaline phosphatase values 1.1 times higher than the upper limit of normal range during screening.
* Volunteers had serum bilirubin value higher than the upper limit of normal range during screening.
* History of bleeding disorders or any significant family history of bleeding disorders.
* History of prosthetic heart valve or history of pulmonary embolism.
* History of traumatic or repeated epidural or spinal puncture or plan for spinal surgery/spinal procedure or volunteer having any spinal deformity or neurological impairment.
* Creatinine clearance below 60 mL/min during screening.
* History or presence of active pathological bleeding.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2024-08-30 (Actual); Primary Completion 2024-10-25 (Actual); Study Completion 2024-11-11 (Actual)

PRIMARY OUTCOMES:
Maximum measured plasma concentration over the time span specified (Cmax) | 36 hours
  acceptance range for 90% confidence interval was considered within 80.00% to 125.00% to establish bioequivalence for Cmax parameter.
The area under the plasma concentration versus time curve was calculated using the linear trapezoidal rule from the zero time point to the last quantifiable concentration (AUCt) | 36 hours
  The 90% confidence interval of the relative mean (Geometric mean) of the Test to reference formulation for Ln-transformed AUCt was to be within 80.00% to 125.00% for Edoxaban to establish bioequivalence

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve to infinity (AUCi) | 36 hours
  Descriptive Statistics
Time of the maximum measured plasma concentration (Tmax) | 36 hours
  Descriptive Statistics

CONTACTS AND LOCATIONS:
Locations (1):
- Cliantha Research Limited, Ahmedabad, Gujarat, India